CLINICAL TRIAL: NCT00006118
Title: First Line Treatment of Locally Advanced or Metastatic Urothelial Carcinoma of the Bladder With a Combination of Cisplatin-Paclitaxel-Gemcitabine
Brief Title: Cisplatin, Paclitaxel, and Gemcitabine in Treating Patients With Progressive Unresectable Regional or Metastatic Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068131; FRE-GERCOR-U99-1; EU-20030
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2001-11

CONDITIONS: Bladder Cancer
Keywords: stage III bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining cisplatin, paclitaxel, and gemcitabine in treating patients who have progressive unresectable regional or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and toxicity of cisplatin, paclitaxel, and gemcitabine in patients with progressive unresectable regional or metastatic transitional cell carcinoma of the bladder.
* Determine the progression free survival of these patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV over 1 hour and paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks for 6 courses.

Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven progressive unresectable regional or metastatic transitional cell carcinoma of the bladder
* Measurable disease by CT or MRI scan

  * Greater than 10 mm

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine less than 1.36 mg/dL

Cardiovascular:

* No uncontrolled cardiac disease
* No severe cardiac arrhythmias

Other:

* Not pregnant or nursing
* No other prior malignancy except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior intravesical immunotherapy for superficial disease allowed
* No prior systemic biologic response modifier therapy for advanced disease

Chemotherapy:

* Prior intravesical chemotherapy for superficial disease allowed
* No prior systemic chemotherapy for advanced disease

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* No prior surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Maulard-Durdux, MD, Study Chair — Hopital Tenon
Locations (12):
- France (11):
  - Hopital Drevon, Dijon
  - CHR de Grenoble - La Tronche, Grenoble
  - Hopital Perpetuel Secours, Levallois-Perret
  - CHU de la Timone, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Laennec, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Tenon, Paris
  - Polyclinique De Courlancy, Reims
  - C.H. Senlis, Senlis
  - Centre Hospitalier Regional Metz Thionville, Thionville
- Centre Hospitalier Princesse Grace, Monte Carlo, Monaco